CLINICAL TRIAL: NCT04415944
Title: A Phase II Trial Evaluating Feasibility and Quality of Life of Second Look Laparoscopy With HIPEC in Patients With Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Trial Evaluating Feasibility and Quality of Life of Second Look Laparoscopy With Hyperthermic Intraperitoneal Chemotherapy
Acronym: HIPEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00066278; WFBCCC 04619 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Epithelial Cancer Stage I; Ovarian Epithelial Cancer Stage II; Ovarian Epithelial Cancer Stage III; Stage I Fallopian Tube Cancer; Stage II Fallopian Tube Cancer; Stage III Fallopian Tube Cancer; Peritoneal Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Second Look Laparoscopy and HIPEC with Carboplatin (Experimental): Laparoscopic assessment of disease status of the peritoneal cavity with lysis of adhesions as necessary noting either no gross residual disease or minimal residual disease prior to or after resection. This is performed prior to establishment of a peritoneal perfusion circuit and hyperthermic intraperitoneal chemotherapy.
  Interventions: Procedure: Second look laparoscopy reassessment surgery (SLLRS); Drug: HIPEC with Carboplatin; Other: FACT-O Quality of Life Questionnaire

INTERVENTIONS:
Procedure: Second look laparoscopy reassessment surgery (SLLRS) — Performed less than 12 weeks after intravenous chemotherapy cycles are completed.
Drug: HIPEC with Carboplatin — Patient receives HIPEC with CBDCA 800 mg/m2 for 90 minutes.
  Patients who exhibit the following will not receive the HIPEC procedure:
  * Extraperitoneal disease noted at the time of the second look procedure
  * Macroscopic intraperitoneal disease which is not resectable to R1
  * Technical problems which prevent continuous, adequate flow to maintain intraperitoneal temperature to 41°C during perfusion
  * Intraoperative complications such as cardiac or pulmonary instability precluding HIPEC
  Participation will consist of completing surveys regarding their cancer and allowing researchers to use information from their medical records for research.
Other: FACT-O Quality of Life Questionnaire — Participants will be asked to do this three times (pre-study, 3 months and 6 months). Surveys will be given at follow up visits for surgery. They should take about 10-15 minutes to complete.

SUMMARY:
The purpose of this research study is to see if it is feasible to receive heated chemotherapy or heated intraperitoneal chemotherapy (HIPEC) inserted directly into the abdomen at the time of a Second Look Reassessment Surgery and to monitor any effects good or bad that this has on participants' health.

DETAILED DESCRIPTION:
Primary Objective: Determine the feasibility of second look laparoscopy and hyperthermic intraperitoneal chemotherapy with carboplatin.

Secondary Objective(s)

* To compare the quality if life in patients with ovarian cancer after undergoing second look laparoscopic reassessment surgery with hyperthermic intraperitoneal chemotherapy using carboplatin (CBDCA) versus quality of life in patients treated with cytoreduction surgery and systemic chemotherapy alone.
* To describe toxicities in patients with ovarian cancer treated with second look laparoscopy and simultaneous hyperthermic intraperitoneal chemotherapy.

OUTLINE:

Patients undergo second look laparoscopy. Patients with visible signs of cancer in abdomen also receive HIPEC with carboplatin via intraperitoneal injection (IP) over 90 minutes in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically I-III epithelial carcinoma of the ovary, fallopian tube or peritoneum or Stage IVA disease in which is there complete resolution of disease (pleural effusion) with chemotherapy
* Patients must have undergone cytoreductive surgery and 3-8 cycles of platinum-based systemic chemotherapy prior to the second look surgery. Systemic platinum based chemotherapy must be completed less than 18 weeks prior to second look surgery.
* Cytoreductive surgery must result in an R-0, R-1 resection prior to systemic chemotherapy
* The intraoperative peritoneal adhesion index should be < 10.
* Patients must be without clinical evidence of disease including a negative exam, imaging (CT or PET/CT) and normal tumor markers (CA125) after completion of systemic chemotherapy.
* Age ≥ 18 years.
* ECOG performance status ≤ 2.
* Patients must have adequate organ and marrow function as defined below (within 30 days of registration): absolute neutrophil count >1,500/mcL; platelets >100,000/mcL; total bilirubin ≤ 1.5 mg/dL; creatinine clearance ≥ 50 mg/dL; AST(SGOT)/ALT(SGPT) ≤ 3X; institutional upper limit of normal; alkaline phosphatase 3X institutional upper limit of normal
* Adequate contraception and negative pregnancy test if pregnancy possible.
* Ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria:

* Patients greater than 18 weeks from their last course of systemic platinum based chemotherapy
* Patients who have received additional chemotherapy for the ovarian cancer after primary therapy as outlined above.
* Patients may not have received prior abdominal or pelvic radiation.
* Extensive intra-abdominal adhesive disease noted at the time of initial cytoreductive surgery with PAI of >10 as defined above
* Intra-abdominal infection associated with initial cytoreductive surgery requiring extended hospitalization or related to systemic chemotherapy requiring hospitalization for therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy

Men are excluded from participation due to the site-specific nature of the disease being studied.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Number of Patients To Successfully Undergo Second Look Laparoscopy and Hyperthermic Intraperitoneal Chemotherapy | Up to 3 months post treatment
  The proportion of feasibility is defined as the number of patients who successfully undergo SLL and HIPEC divided by the number of patients who are eligible and consent to participate. The feasibility proportion and its 95% confidence interval will be estimated.

SECONDARY OUTCOMES:
Quality of Life - Functional Assessment of Cancer Therapy-Ovarian (FACT-O) Questionnaire | Up to 6 months post-treatment
  The quality of life in patients with advanced ovarian cancer after undergoing second look laparoscopy reassessment surgery with hyperthermic intraperitoneal chemotherapy using Carboplatin (CBDCA) will be determined by the FACT-O questionnaire at pre-study, and months 3, and 6 in follow-up (post-treatment). The distribution of quality of life at each visit and the distribution of change in quality of life at each follow-up visit will be examined and the descriptive statistics will be presented. Scoring scale - (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, and 4 = very much) and includes questions relating to Physical Well-Being (7 items), Social Well-being (7 items), Functional Well-Being (7 items), Emotional Well-Being (6 items) and Additional Ovarian Cancer Concerns (12-item). Scores could range from 0-156. Higher scores are associated with better QOL.
Number of Reported Toxicities | Up to 3 months post treatment
  Toxicities will be indicated by the number and severity of adverse events as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. . Counts and percentages will be calculated for each adverse event. Mean, standard deviation, median, and interquartile range will be calculated for number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Berry, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No